CLINICAL TRIAL: NCT06501781
Title: Peer Behavioral Activation Utilization to Improve Substance Use and HIV Outcomes in People Receiving Long Acting Injectable-PrEP/ART (PUSH)
Acronym: PUSH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Elana Rosenthal, Associate Professor MD, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HP-00110311
Record Dates: First submitted 2024-07-02; First posted 2024-07-15 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: HIV Infections; Substance Use
MeSH Terms: conditions — HIV Infections; Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: A pilot study to evaluate the feasibility and effectiveness of a peer-delivered intervention for LAI-PrEP/ART adherence among predominately Black substance-using populations.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Peer Activate-LAI (Experimental): Peer Activate-LAI, is a peer recovery specialist-delivered (PRS) behavioral activation (BA) and problem solving intervention aimed at improving adherence to LAI-PrEP/ART. BA was originally developed as an efficacious treatment for depression, with accumulating empirical support for SUD outcomes, including SUD treatment retention and HIV medication adherence, particularly when integrated with problem solving strategies. BA offers important advantages compared to other psychosocial interventions by being feasible and potentially sustainable for PRS delivery, appropriate for low-income individuals with OUD and other non-opioid SUD, and focused on building positive reinforcement in the current environment through engagement in adaptive, valued behaviors.
  Interventions: Behavioral: Peer Activate-LAI; Other: Standard of Care HIV treatment or prevention with LAI-PrEP/ART
- Enhanced Treatment As Usual (Active Comparator): Participants in the Enhanced Treatment As Usual (ETAU) arm receive access to standard clinical care, including access to a clinician with expertise in HIV and PrEP, opportunity for co-located treatment of OUD, and STI testing and treatment, and general peer support. Enhanced treatment includes reminder phone calls and facilitated referrals to psychosocial, housing, financial benefits and legal services.
  Interventions: Other: Standard of Care HIV treatment or prevention with LAI-PrEP/ART

INTERVENTIONS:
Behavioral: Peer Activate-LAI — Peer Activate-LAI is a Peer Recovery Specialist-delivered behavioral activation and problem solving intervention, based on our team's formative work. The intervention focuses on problem-solving skills to improve adherence to ART and/or PrEP both at the individual level and environmental barriers to care (i.e., transportation, housing).
  Arms: Peer Activate-LAI
Other: Standard of Care HIV treatment or prevention with LAI-PrEP/ART — Standard of care HIV treatment or prevention with LAI-PrEP/ART

SUMMARY:
This randomized Type 1 hybrid effectiveness-implementation trial (N=186) will evaluate the effectiveness and implementation of a peer-delivered problem solving and behavioral activation intervention for adherence to LAI-PrEP/ART ("Peer Activate-LAI") compared to enhanced treatment as usual (ETAU) for a largely Black, substance-using population living with or at high risk for HIV. Specific aims are to:

Aim 1: Evaluate the effectiveness of Peer Activate-LAI over 12-months on: a) LAI-PrEP/ART adherence (primary; receipt of all 6 maintenance injections within 7-day window); and b) substance use (secondary; WHOASSIST, urine toxicology); and c) Explore the moderating role of SRD-related factors (exploratory)

Aim 2: To evaluate the implementation of Peer Activate-LAI including feasibility, acceptability, fidelity, and adoption guided by RE-AIM and Proctor's model,12,13 assessed using mixed methods, including a rapid ethnographic assessment of how SRD-related factors may affect implementation.

Aim 3: To evaluate the economic viability of Peer Activate-LAI, including a) cost of implementation and sustainment, and b) cost-effectiveness from multiple stakeholder perspectives.

This study will inform a potentially scalable, cost-effective model for facilitating effective adherence to LAI formulations of PrEP/ART within Black, substance-using populations with multiple minority identities who to date have had limited support for improving LAI adherence for HIV treatment and prevention.

DETAILED DESCRIPTION:
Background. Substance use continues to be a major driver of HIV acquisition and has been associated with suboptimal ART adherence, treatment interruption, and inability to achieve or maintain viral suppression. Use of PrEP, a key tool for HIV prevention, is disproportionately lower in racial/ethnic minorities, as well as people who inject drugs. Factors related to structural racism and discrimination (SRD) may contribute to low rates of adherence in these populations. New long-acting injectable (LAI) formulations of PrEP/ART provide a potential biomedical intervention to overcome adherence challenges, however, due to the prolonged subtherapeutic period after LAI discontinuation, ensuring adherence is crucial.

A peer-delivered reinforcement-based intervention may be a promising solution for improving LAI adherence. Our team has developed through several rounds of stakeholder feedback a peer-delivered behavioral activation and problem-solving intervention, Peer Activate. Peer Activate focuses on problem-solving skills to improve adherence to ART and/or PrEP both at the individual level and social/structural barriers to care (i.e., transportation, housing) and includes behavioral activation to promote engagement in rewarding, substance-free activities in one's environment and structured daily activities to promote treatment adherence. Delivery by a peer with formal training and shared lived experiences enhances the impact of the intervention on SRD-related factors. However, Peer Activate has not been evaluated in the context of LAI PrEP/ART.

Preliminary Studies. This proposal builds upon our team's prior studies demonstrating 1) our ability to engage patients with and at risk for HIV, facing multiple barriers due to SRD, and provide LAI PrEP/ART in community-based settings; 2) the feasibility and acceptability of Peer Activate and promise in improving HIV treatment adherence for people who use substances.; and 3) promise for cost-effectiveness.

Approach. We propose a randomized Type 1 hybrid effectiveness-implementation trial (N=186) to test the effectiveness and implementation of Peer Activate for LAI PrEP/ART ("Peer Activate-LAI") vs. enhanced treatment as usual for a predominantly Black substance using population living with or at high risk for HIV, evaluating the following over 12 months:

1. effectiveness: a) LAI PrEP/ART adherence (primary; receipt of all 6 maintenance injections within 7-day window); b) substance use (secondary; urine toxicology, self-report); c) SRD as moderators of effectiveness (exploratory);
2. Implementation of Peer Activate-LAI including feasibility, acceptability, fidelity, and adoption guided by RE-AIM and Proctor's model,9,10 assessed using mixed methods, including a rapid ethnographic assessment of how SRD-related factors may affect implementation; and
3. Economic viability of Peer Activate-LAI, including cost of implementation and sustainment and cost-effectiveness from multiple stakeholder perspectives. Implications.

This study will inform a potentially scalable, cost-effective model for facilitating effective adherence to LAI formulations of ART/PrEP within Black, substance using populations who to date have had limited support for improving LAI adherence for HIV ART/PrEP.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Able and willing to sign informed consent
* HIV status:

HIV negative with a negative HIV antibody/antigen test and meeting CDC(center for disease control and prevention) criteria for PrEP HIV positive with a positive antibody/antigen test

* Meeting indications for treatment based on Cabotegravir-LA (HIV negative) or Cabotegravir (CAB) and Rilpivirine (RPV)-LA (HIV positive) prescribing information
* Moderate substance use, defined as a (World Health Organization Alcohol, Smoking and Substance Involvement Screening Test) WHO-ASSIST score of ≥4 for certain drugs (cocaine, amphetamines, inhalants, sedatives, hallucinogens, or opioids) or ≥11 for alcohol

Exclusion Criteria:

* Contraindications to Cabotegravir-LA (HIV-) or Cabotegravir (CAB) and Rilpivirine (RPV)-LA (HIV+) use based on prescribing information or other medical/psychiatric conditions that may interfere with study participation
* Pregnant or breastfeeding

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
LAI-PrEP/ART Complete Adherence | 12 months
  Defined as receiving all 6 LAI maintenance doses within the +/-7 day window.
  Unit of Measure: Binary (Yes/No)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - HIPS (Harm reduction drop-in center), Washington D.C., District of Columbia
  - Baltimore Safe Haven, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No